CLINICAL TRIAL: NCT04221945
Title: A Randomized, Phase 3, Double-Blind Study of Chemoradiotherapy With or Without Pembrolizumab for the Treatment of High-risk, Locally Advanced Cervical Cancer (KEYNOTE-A18/ENGOT-cx11/GOG-3047)
Brief Title: Study of Chemoradiotherapy With or Without Pembrolizumab (MK-3475) For The Treatment of Locally Advanced Cervical Cancer (MK-3475-A18/KEYNOTE-A18/ENGOT-cx11/GOG-3047)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: GOG Foundation (Network); European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3475-A18; MK-3475-A18 (Other: MSD); KEYNOTE-A18 (Other: MSD); ENGOT-cx11 (Other: European Network for Gynaecological Oncological Trial groups); 205189 (Registry Identifier: JAPAC-CTI); GOG-3047 (Other: Gynecologic Oncology Group Foundation); 2022-501972-25-00 (Registry Identifier: EU CT); U1111-1282-6395 (Registry Identifier: UTN); 2019-003152-37 (EudraCT Number)
Record Dates: First submitted 2019-12-23; First posted 2020-01-09 (Actual); Results first posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Programmed Cell Death Receptor 1 (PD-1, PD1); Programmed Cell Death Receptor Ligand 1 (PD-L1, PDL1); Programmed Cell Death Receptor Ligand 2 (PD-L2, PDL2)
MeSH Terms: conditions — Uterine Cervical Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Cisplatin; Brachytherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- chemoradiotherapy + pembrolizumab (Experimental): Participants receive pembrolizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle (Q3W) for 5 cycles followed by pembrolizumab 400 mg IV on Day 1 of each 6-week cycle (Q6W) for an additional 15 cycles. During the Q3W dosing period of pembrolizumab, participants receive concurrent chemoradiotherapy. The standard of care chemoradiotherapy regimen includes cisplatin 40 mg/m^2 IV once per week (QW) for 5 or 6 weeks plus external beam radiotherapy (EBRT) followed by brachytherapy with minimum total radiotherapy dose of 80 Gray Units (Gy) for volume-directed and 75 Gy for point-directed given with the total duration of radiation treatment not to exceed 50 days (with an extension to a maximum of 56 days for unforeseen delays).
  Interventions: Biological: Pembrolizumab; Drug: Cisplatin; Radiation: External Beam Radiotherapy (EBRT); Radiation: Brachytherapy
- chemoradiotherapy + placebo for pembrolizumab (Experimental): Participants receive placebo for pembrolizumab IV on Day 1 of each 3-week cycle (Q3W) for 5 cycles followed by placebo IV on Day 1 of each 6-week cycle (Q6W) for an additional 15 cycles. During the Q3W dosing period of placebo, participants receive concurrent chemoradiotherapy. The standard of care chemoradiotherapy regimen includes cisplatin 40 mg/m^2 IV once per week (QW) for 5 or 6 weeks plus external beam radiotherapy (EBRT) followed by brachytherapy with minimum total radiotherapy dose of 80 Gray Units (Gy) for volume-directed and 75 Gy for point-directed given with the total duration of radiation treatment not to exceed 50 days (with an extension to a maximum of 56 days for unforeseen delays).
  Interventions: Drug: Placebo for pembrolizumab; Drug: Cisplatin; Radiation: External Beam Radiotherapy (EBRT); Radiation: Brachytherapy

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: KEYTRUDA®; MK-3475
  Arms: chemoradiotherapy + pembrolizumab
Drug: Placebo for pembrolizumab — IV infusion
  Arms: chemoradiotherapy + placebo for pembrolizumab
Drug: Cisplatin — IV infusion
  Other Names: Platinol®; Platinol®-AQ
Radiation: External Beam Radiotherapy (EBRT) — Given as a total radiotherapy dose of 80 Gy for volume-directed and 75 Gy for point-directed
Radiation: Brachytherapy — Given as a total radiotherapy dose of 80 Gy for volume-directed and 75 Gy for point-directed

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of pembrolizumab plus concurrent chemoradiotherapy compared to placebo plus concurrent chemoradiotherapy in participants with locally advanced cervical cancer.

The primary hypotheses are that pembrolizumab plus concurrent chemoradiotherapy is superior to placebo plus concurrent chemoradiotherapy with respect to progression-free survival and overall survival.

Once the study objectives have been met or the study has ended, participants will be discontinued from this study and will be enrolled in an extension study to continue protocol-defined assessments and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Has high-risk locally advanced cervical cancer (LACC): The International Federation of Gynecology and Obstetrics (FIGO) 2014 Stage IB2-IIB (with node-positive disease) or FIGO 2014 Stages III-IVA
* Has histologically-confirmed squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma of the cervix
* Has not previously received any definitive surgical, radiation, or systemic therapy for cervical cancer, including investigational agents, and is immunotherapy-naïve
* Female participants must not be pregnant or breastfeeding and agree to use highly effective contraception during the treatment period and for at least 120 days after the last dose of pembrolizumab or placebo and 180 days following the end of chemoradiotherapy and agrees not to donate eggs (ova, oocytes) to others or freeze/store for her own use for the purpose of reproduction during this period.
* Female participants must abstain from breastfeeding during the study intervention period and for at least 120 days after the last dose of pembrolizumab or placebo and 180 days following the end of chemoradiotherapy
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 7 days prior to the first dose of study treatment
* Has provided a tissue sample from a core incisional or excisional biopsy of a tumor lesion
* Has radiographically evaluable disease, either measurable or non-measurable per RECIST 1.1, as assessed by the local site investigator/radiology
* Has adequate organ function within 7 days prior to the start of study treatment.

Exclusion Criteria:

* Has excluded subtypes of LACC
* Has FIGO 2014 Stage IVB disease
* Has undergone a previous hysterectomy defined as removal of the entire uterus or will have a hysterectomy as part of their initial cervical cancer therapy
* Has bilateral hydronephrosis, unless at least one side has been stented or resolved by positioning of nephrostomy or considered mild and not clinically significant in the opinion of the investigator
* Has anatomy or tumor geometry or any other reason or contraindication that cannot be treated with intracavitary brachytherapy or a combination of intracavitary and interstitial brachytherapy
* Has received a live vaccine within 30 days prior to the first dose of study treatment
* Has received treatment with systemic immunostimulatory agents, colony stimulating factors, interferons, interleukins and vaccine combinations within 6 weeks or 5 half-lives of the drug, whichever is shorter, prior to Cycle 1, Day 1
* Has received prior therapy with an anti-programmed cell death receptor 1 (PD-1), anti-programmed cell death receptor ligand 1 (PD-L1), or anti-programmed cell death receptor ligand 2 (PD-L2) agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), OX-40, CD137)
* Has received prior systemic anticancer therapy including investigational agents within 4 weeks prior to randomization
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to randomization
* Has any contraindication to the use of cisplatin
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has severe hypersensitivity to pembrolizumab and/or any of its excipients
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy
* Has a known history of Human Immunodeficiency Virus (HIV) infection
* Has a known history of Hepatitis B or known active Hepatitis C virus infection
* Has a history or current evidence of any condition, therapy, lab abnormality, or other circumstance that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results, and in the judgment of the investigator or Sponsor, would make the participant inappropriate for entry into this study
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study
* Has had an allogenic tissue/solid organ transplant
* Has evidence of metastatic disease per RECIST 1.1 including lymph nodes above the first lumbar vertebra (L1) cephalad body, in the inguinal region

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1060 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2026-01-17 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (176):
- United States (28):
  - HonorHealth Research Institute - Biltmore ( Site 8009), Phoenix, Arizona
  - UCLA Hematology/Oncology - Westwood (Building 200 Suite 120) ( Site 0027), Los Angeles, California
  - Hoag Memorial Hospital Presbyterian ( Site 0038), Newport Beach, California
  - UC Davis Comprehensive Cancer Center ( Site 0017), Sacramento, California
  - University of Colorado Health Sciences Center and Hospital ( Site 0028), Denver, Colorado
  - Smilow Cancer Center at Yale-New Haven ( Site 0023), New Haven, Connecticut
  - AdventHealth Orlando-AdventHealth Medical Group Gynecological Oncology ( Site 0009), Orlando, Florida
  - Parkview Research Center at Parkview Regional Medical Center ( Site 0026), Fort Wayne, Indiana
  - University of Kentucky Markey Cancer Center ( Site 0015), Lexington, Kentucky
  - Our Lady of the Lake Regional Medical Center. ( Site 0031), Baton Rouge, Louisiana
  - Women's Cancer Care ( Site 0039), Covington, Louisiana
  - Karmanos Cancer Institute ( Site 0018), Detroit, Michigan
  - Minnesota Oncology Hematology, PA ( Site 8007), Minneapolis, Minnesota
  - University of New Mexico Comprehensive Cancer Center-Clinical Research Office ( Site 0019), Albuquerque, New Mexico
  - University of North Carolina at Chapel Hill ( Site 0025), Chapel Hill, North Carolina
  - Sanford Bismarck Medical Center ( Site 0046), Bismarck, North Dakota
  - The James Cancer Hospital and Solove Research Institute at The Ohio State University Comprehensive C, Columbus, Ohio
  - Willamette Valley Cancer Institute and Research Center ( Site 8000), Eugene, Oregon
  - Legacy Good Samaritan Medical Center ( Site 0013), Portland, Oregon
  - Allegheny Health Network West Penn Hospital-Gynecologic Oncology ( Site 0030), Pittsburgh, Pennsylvania
  - Hollings Cancer Center ( Site 0007), Charleston, South Carolina
  - Sanford Gynecology Oncology ( Site 0003), Sioux Falls, South Dakota
  - Texas Oncology-Austin Central ( Site 8006), Austin, Texas
  - Texas Oncology-Fort Worth Cancer Center ( Site 8001), Fort Worth, Texas
  - Texas Oncology-San Antonio Medical Center ( Site 8002), San Antonio, Texas
  - Texas Oncology-The Woodlands ( Site 8003), The Woodlands, Texas
  - UVA Health System ( Site 0005), Charlottesville, Virginia
  - Virginia Commonwealth University ( Site 0024), Richmond, Virginia
- Australia (5):
  - Westmead Hospital ( Site 0973), Westmead, New South Wales
  - Royal Brisbane and Women s Hospital ( Site 0972), Herston, Queensland
  - Monash Health-Monash Medical Centre ( Site 0970), Clayton, Victoria
  - Peter MacCallum Cancer Centre ( Site 0971), Melbourne, Victoria
  - St John of God Subiaco Hospital ( Site 0969), Subiaco, Western Australia
- Austria (3):
  - Medizinische Universitat Graz ( Site 0569), Graz, Styria
  - Medizinische Universitat Innsbruck ( Site 0566), Innsbruck, Tyrol
  - Medizinische Universität Wien ( Site 0567), Vienna, Vienna
- Belgium (6):
  - UZA University Hospital Antwerp ( Site 0351), Edegem, Antwerpen
  - GZA Sint Augustinus ( Site 0356), Wilrijk, Antwerpen
  - C.I.U. Hopital Ambroise Pare ( Site 0353), Mons, Hainaut
  - OLV Ziekenhuis ( Site 0352), Aalst, Oost-Vlaanderen
  - AZ St Lucas ( Site 0349), Ghent, Oost-Vlaanderen
  - UZ Leuven ( Site 0354), Leuven, Vlaams-Brabant
- Brazil (5):
  - Hospital das Clinicas da UFMG ( Site 0172), Belo Horizonte, Minas Gerais
  - Liga Norte Riograndense Contra o Cancer ( Site 0170), Natal, Rio Grande do Norte
  - Hospital de Clínicas de Ribeirão Preto ( Site 0171), Ribeirão Preto, São Paulo
  - Núcleo de Pesquisa Clínica da Rede São Camilo ( Site 0166), São Paulo, São Paulo
  - Instituto Nacional Do Cancer II ( Site 0173), Rio de Janeiro
- Canada (4):
  - Princess Margaret Cancer Centre ( Site 0102), Toronto, Ontario
  - Centre Hospitalier de l Universite de Montreal - CHUM ( Site 0101), Montreal, Quebec
  - McGill University Health Centre ( Site 0105), Montreal, Quebec
  - Centre intégré de cancérologie du CHU de Québec Université Laval, Hôpital de l'Enfant-Jésus ( Site 0, Québec, Quebec
- Chile (4):
  - Sociedad Oncovida S.A. ( Site 0196), Santiago, Region M. de Santiago
  - Iram Cancer Research ( Site 0198), Santiago, Region M. de Santiago
  - Centro Investigación del Cáncer James Lind ( Site 0194), Temuco, Región de la Araucanía
  - Oncocentro ( Site 0195), Viña del Mar, Región de Valparaíso
- China (16):
  - Anhui Provincial Hospital ( Site 1029), Hefei, Anhui
  - Anhui Provincial Cancer Hospital ( Site 1007), Hefei, Anhui
  - Peking Union Medical College Hospital ( Site 1001), Beijing, Beijing Municipality
  - Chongqing Cancer Hospital ( Site 1030), Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University ( Site 1025), Xiamen, Fujian
  - The First Affiliated Hospital.Sun Yat-sen University ( Site 1005), Guangzhou, Guangdong
  - Affiliated Cancer Hospital of Guangxi Medical University ( Site 1036), Nanning, Guangxi
  - Harbin Medical University Cancer Hospital ( Site 1013), Harbin, Heilongjiang
  - Hunan Cancer Hospital ( Site 1015), Changsha, Hunan
  - Xiangya Hospital Central-South University ( Site 1009), Changsha, Hunan
  - Shanghai Cancer Hospital ( Site 1000), Shanghai, Shanghai Municipality
  - Shanghai First Maternity and Infant Hospital-Gynecology department ( Site 1039), Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital ( Site 1018), Chengdu, Sichuan
  - The First Affiliated Hospital of Xinjiang Medical University ( Site 1012), Ürümqi, Xinjiang
  - Zhejiang Provincial People's Hospital ( Site 1021), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 1004), Hangzhou, Zhejiang
- Colombia (4):
  - Fundacion Centro de Investigacion Clinica CIC ( Site 0231), Medellín, Antioquia
  - Instituto Nacional de Cancerologia E.S.E ( Site 0228), Bogotá, Bogota D.C.
  - Fundacion Valle del Lili ( Site 0230), Cali, Valle del Cauca Department
  - Centro Medico Imbanaco de Cali S.A ( Site 0227), Cali, Valle del Cauca Department
- Czechia (3):
  - Fakultni Nemocnice Brno Bohunice ( Site 0912), Brno, Brno-mesto
  - Fakultni nemocnice Ostrava ( Site 0909), Ostrava, Moravskoslezský kraj
  - Fakultni nemocnice Kralovske Vinohrady ( Site 0913), Prague
- France (3):
  - CHU Jean Minjoz ( Site 0411), Besançon, Doubs
  - Institut Claudius Regaud ( Site 0417), Toulouse, Haute-Garonne
  - Centre Hospitalier Lyon Sud ( Site 0413), Pierre-Bénite, Rhone
- Germany (8):
  - Universitaetsklinikum Freiburg ( Site 0454), Freiburg im Breisgau, Baden-Wurttemberg
  - Universitätsmedizin Mannheim-Department of Obstetrics and Gynecology ( Site 0443), Mannheim, Baden-Wurttemberg
  - Klinikum der Universitaet in Muenchen ( Site 0446), Munich, Bavaria
  - Klinikum Rechts der Isar. Technischen Universitaet Muenchen ( Site 0453), Munich, Bavaria
  - Universitaetsklinikum Carl Gustav Carus der Technischen Univ ( Site 0452), Dresden, Saxony
  - Universitaetsklinik Leipzig ( Site 0456), Leipzig, Saxony
  - Charite Universitaetsmedizin Berlin ( Site 0442), Berlin
  - Universitaetsklinikum Hamburg-Eppendorf ( Site 0445), Hamburg
- Greece (4):
  - General Hospital of Patras. St Andrews ( Site 0473), Pátrai, Achaia
  - Alexandra General Hospital ( Site 0477), Athens, Attica
  - Hospital Hygeia ( Site 0478), Athens, Attica
  - Euromedica General Clinic of Thessaloniki ( Site 0474), Thessaloniki
- Guatemala (6):
  - Centro de Investigaciones Clinicas de Latinoamerica S.A. - CELAN ( Site 0321), Guatemala City
  - Oncologika S.A. ( Site 0323), Guatemala City
  - Oncomedica ( Site 0320), Guatemala City
  - Grupo Angeles SA ( Site 0319), Guatemala City
  - Medi-K Cayala ( Site 0318), Guatemala City
  - Centro Medico Integral De Cancerología (CEMIC) ( Site 0322), Quetzaltenango
- Hungary (2):
  - Orszagos Onkologiai Intezet ( Site 0846), Budapest
  - Debreceni Egyetem Klinikai Kozpont ( Site 0845), Debrecen
- Ireland (2):
  - Cork University Hospital ( Site 0504), Cork
  - St James Hospital ( Site 0505), Dublin
- Israel (4):
  - Rambam Medical Center ( Site 0815), Haifa
  - Hadassah Medical Center. Ein Kerem ( Site 0816), Jerusalem
  - Chaim Sheba Medical Center ( Site 0814), Ramat Gan
  - Sourasky Medical Center ( Site 0819), Tel Aviv
- Italy (10):
  - Istituto Europeo di Oncologia ( Site 0536), Milan, Milano
  - Istituto di Candiolo - IRCCS ( Site 0546), Candiolo, Piedmont
  - Istituto Nazionale Tumori Regina Elena ( Site 0540), Rome, Roma
  - A.O. Universitaria Policlinico S. Orsola-Malpighi ( Site 0541), Bologna
  - Ospedale Vito Fazzi ( Site 0547), Lecce
  - IRCCS Ospedale San Raffaele ( Site 0539), Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano ( Site 0542), Milan
  - Fondazione Giovanni Pascale Di Napoli ( Site 0544), Napoli
  - Policlinico Universitario Gemelli ( Site 0538), Roma
  - A.O.U. Citta della Salute e della Scienza di Torino ( Site 0535), Torino
- Japan (17):
  - Aichi Cancer Center Hospital ( Site 1155), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 1159), Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center ( Site 1162), Matsuyama, Ehime
  - Ehime University Hospital ( Site 1157), Tōon, Ehime
  - Kurume University Hospital ( Site 1164), Kurume, Fukuoka
  - Hokkaido University Hospital ( Site 1163), Sapporo, Hokkaido
  - Iwate Medical University Hospital ( Site 1165), Shiwa-gun, Iwate
  - University of the Ryukyus Hospital ( Site 1156), Nakagami-gun, Okinawa
  - Saitama Medical University International Medical Center ( Site 1168), Hidaka, Saitama
  - Saitama Cancer Center ( Site 1169), Kitaadachi-gun, Saitama
  - Kyorin University Hospital ( Site 1158), Mitaka, Tokyo
  - National Hospital Organization Kyushu Cancer Center ( Site 1167), Fukuoka
  - Kagoshima City Hospital ( Site 1166), Kagoshima
  - Osaka International Cancer Institute ( Site 1161), Osaka
  - National Cancer Center Hospital ( Site 1172), Tokyo
  - Japanese Foundation for Cancer Research-Gynecologic Oncology ( Site 1171), Tokyo
  - Keio University Hospital ( Site 1170), Tokyo
- Norway (2):
  - Helse Bergen HF Haukeland Universitetssjukehus ( Site 0601), Bergen, Hordaland
  - Oslo Universitetssykehus Radiumhospitalet ( Site 0600), Oslo
- Peru (7):
  - Centro Medico Monte Carmelo ( Site 0289), Arequipa, Ariqipa
  - Hospital de Alta Complejidad de La Libertad Virgen de La Puerta ( Site 0287), Trujillo, La Libertad
  - Clinica San Gabriel ( Site 0296), San Miguel, Lima region
  - Hospital Nacional Daniel Alcides Carrion ( Site 0293), Callao, Lima
  - Instituto de Oncologia y Radioterapia Clinica Ricardo Palma ( Site 0290), Lima
  - Hospital Nacional Arzobispo Loayza ( Site 0292), Lima
  - Hospital Nacional Guillermo Almenara Irigoyen ( Site 0291), Lima
- Russia (6):
  - Chelyabinsk Regional Clinical Center Oncology and Nuclear Medicine ( Site 0741), Chelyabinsk, Chelyabinsk Oblast
  - Krasnoyarsk Regional Clinical Oncological Dispensary ( Site 0729), Krasnoyarsk, Krasnoyarsk Krai
  - MSROI named after P.A. Hertsen branch of FSBI NMRC Radiology ( Site 0722), Moscow, Moscow
  - GBUZ SPb CRPCstmc(o) ( Site 0746), Saint Petersburg, Sankt-Peterburg
  - National Medical Research Center of Oncology N.A. N.N. Petrov ( Site 0725), Saint Petersburg, Sankt-Peterburg
  - Yaroslavl Regional SBIH Clinical Oncology Hospital ( Site 0734), Yaroslavl, Yaroslavl Oblast
- South Korea (5):
  - National Cancer Center ( Site 1065), Goyang-si, Kyonggi-do
  - Asan Medical Center ( Site 1062), Seoul, Seoul
  - Keimyung University Dongsan Medical Center ( Site 1066), Daegu, Taegu-Kwangyokshi
  - Severance Hospital ( Site 1063), Seoul
  - Samsung Medical Center ( Site 1064), Seoul
- Spain (6):
  - Hospital Germans Trias i Pujol-Instituto Catalán de Oncología de Badalona ( Site 0637), Badalona, Barcelona
  - Hosp Clin Univ de Santiago ( Site 0629), Santiago de Compostela, La Coruna
  - HOSPITAL UNIVERSITARIO QUIRONSALUD MADRID-ONCOLOGIA MEDICA ( Site 0638), Pozuelo de Alarcón, Madrid
  - Hospital Universitari Vall d Hebron ( Site 0634), Barcelona
  - Complejo Hospitalario de Jaen ( Site 0632), Jaén
  - Hospital Clinico Universitario Lozano Blesa ( Site 0630), Zaragoza
- Karolinska Universitetssjukhuset ( Site 0784), Stockholm, Stockholm County, Sweden
- Taiwan (3):
  - National Taiwan University Hospital ( Site 1095), Taipei
  - Mackay Memorial Hospital ( Site 1094), Taipei
  - Linkou Chang Gung Memorial Hospital ( Site 1097), Taoyuan District
- Thailand (4):
  - Ramathibodi Hospital, Mahidol University ( Site 1131), Rajthevee, Bangkok
  - Srinagarind Hospital. Khon Kaen University ( Site 1132), Mueang, Changwat Khon Kaen
  - Songklanagarind Hospital ( Site 1130), Hat Yai, Changwat Songkhla
  - Maharaj Nakorn Chiang Mai Hospital ( Site 1133), Chiang Mai
- Turkey (Türkiye) (3):
  - I.U. Cerrahpasa Medical Faculty ( Site 0755), Istanbul, Istanbul
  - Acibadem Adana Hastanesi ( Site 0756), Adana
  - Baskent Universitesi Ankara Hastanesi ( Site 0754), Ankara
- Ukraine (2):
  - Grigoriev Institute for medical Radiology NAMS of Ukraine ( Site 0876), Kharkiv, Kharkivs’ka Oblast’
  - Lviv State Oncology Regional Treatment and Diagnostic Center ( Site 0882), Lviv, Lviv Oblast
- United Kingdom (3):
  - Royal Devon and Exeter Foundation Trust Hospital ( Site 0699), Exeter, England
  - ROYAL MARSDEN HOSPITAL (CHELSEA) ( Site 0701), London, London, City of
  - Royal Marsden Hospital (Sutton)-Gynaecology Unit ( Site 0696), London, Surrey

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Lorusso D, Xiang Y, Hasegawa K, Scambia G, Leiva M, Ramos-Elias P, Acevedo A, Sukhin V, Cloven N, Pereira de Santana Gomes AJ, Contreras Mejia F, Reiss A, Ayhan A, Lee JY, Saevets V, Zagouri F, Gilbert L, Sehouli J, Tharavichitkul E, Lindemann K, Lazzari R, Chang CL, Lampe R, Zhu H, Oaknin A, Christiaens M, Polterauer S, Usami T, Li K, Yamada K, Toker S, Keefe SM, Pignata S, Duska LR; ENGOT-cx11/GOG-3047/KEYNOTE-A18 investigators. Pembrolizumab or placebo with chemoradiotherapy followed by pembrolizumab or placebo for newly diagnosed, high-risk, locally advanced cervical cancer (ENGOT-cx11/GOG-3047/KEYNOTE-A18): a randomised, double-blind, phase 3 clinical trial. Lancet. 2024 Apr 6;403(10434):1341-1350. doi: 10.1016/S0140-6736(24)00317-9. Epub 2024 Mar 20. PMID 38521086
- [Result] Lorusso D, Xiang Y, Hasegawa K, Scambia G, Leiva M, Ramos-Elias P, Acevedo A, Cvek J, Randall L, Pereira de Santana Gomes AJ, Contreras Mejia F, Helpman L, Akilli H, Lee JY, Saevets V, Zagouri F, Gilbert L, Sehouli J, Tharavichitkul E, Lindemann K, Colombo N, Chang CL, Bednarikova M, Zhu H, Oaknin A, Christiaens M, Petru E, Usami T, Liu P, Yamada K, Toker S, Keefe SM, Pignata S, Duska LR; ENGOT-cx11/GOG-3047/KEYNOTE-A18 investigators. Pembrolizumab or placebo with chemoradiotherapy followed by pembrolizumab or placebo for newly diagnosed, high-risk, locally advanced cervical cancer (ENGOT-cx11/GOG-3047/KEYNOTE-A18): overall survival results from a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2024 Oct 5;404(10460):1321-1332. doi: 10.1016/S0140-6736(24)01808-7. Epub 2024 Sep 14. PMID 39288779
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26324&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The following participants were enrolled: had high-risk IB2-IIB (node-positive) or Stage III-IVA locally advanced cervical cancer (LACC); had histologically confirmed squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma of the cervix; had not previously received any definitive surgical, radiation, or systemic therapy for cervical cancer, including investigational agents, and was immunotherapy-naïve; had an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
Groups:
- Chemoradiotherapy + Pembrolizumab: Participants received pembrolizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle (Q3W) for 5 cycles followed by pembrolizumab 400 mg IV on Day 1 of each 6-week cycle (Q6W) for an additional 15 cycles. During the Q3W dosing period of pembrolizumab, participants received concurrent chemoradiotherapy. The standard of care chemoradiotherapy regimen includes cisplatin 40 mg/m^2 IV once per week (QW) for 5 or 6 weeks plus external beam radiotherapy (EBRT) followed by brachytherapy with minimum total radiotherapy dose of 80 Gray Units (Gy) for volume-directed and 75 Gy for point-directed given with the total duration of radiation treatment not to exceed 50 days (with an extension to a maximum of 56 days for unforeseen delays).
- Chemoradiotherapy + Placebo for Pembrolizumab: Participants received placebo for pembrolizumab IV on Day 1 of each 3-week cycle (Q3W) for 5 cycles followed by placebo IV on Day 1 of each 6-week cycle (Q6W) for an additional 15 cycles. During the Q3W dosing period of placebo, participants received concurrent chemoradiotherapy. The standard of care chemoradiotherapy regimen includes cisplatin 40 mg/m^2 IV once per week (QW) for 5 or 6 weeks plus external beam radiotherapy (EBRT) followed by brachytherapy with minimum total radiotherapy dose of 80 Gray Units (Gy) for volume-directed and 75 Gy for point-directed given with the total duration of radiation treatment not to exceed 50 days (with an extension to a maximum of 56 days for unforeseen delays).
Period: Overall Study
Arm/Group | Chemoradiotherapy + Pembrolizumab | Chemoradiotherapy + Placebo for Pembrolizumab
Started (Randomized) | 529 | 531
Treated | 528 | 530
Completed | 0 | 0
Not Completed | 529 | 531
Not completed — Death | 103 | 140
Not completed — Lost to Follow-up | 5 | 8
Not completed — Withdrawal by Subject | 21 | 11
Not completed — Participants Ongoing | 400 | 372

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemoradiotherapy + Pembrolizumab | Chemoradiotherapy + Placebo for Pembrolizumab | Total
Number analyzed (Participants) | 529 | 531 | 1060
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.4 (11.9) | 50.1 (12.3) | 49.8 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 529 | 531 | 1060
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 161 | 173 | 334
  Not Hispanic or Latino | 363 | 356 | 719
  Unknown or Not Reported | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 24 | 22 | 46
  Asian | 156 | 148 | 304
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 14 | 8 | 22
  White | 254 | 264 | 518
  More than one race | 78 | 86 | 164
  Unknown or Not Reported | 1 | 2 | 3
PDL-1 Status [Count of Participants; unit: Participants] — Programmed cell death ligand 1 (PDL-1) status based on combined positive score (CPS) indicates tumor PD-L1 positivity using both tumor cells and inflammatory cells that are positive for PD-L1 by IHC. The number of participants with CPS<1 and CPS ≥1 at baseline is presented. Participants with CS <1 were classified as PD-L1 negative, and participants with CPS ≥1 were classified as PD-L1 positive.
  Participants
    CPS<1 | 22 | 28 | 50
    CPS>=1 | 502 | 498 | 1000
    Missing | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by the Investigator
Description: PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, or by histopathologic confirmation of suspected disease progression, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. Unequivocal progression of non-target lesions is also considered PD. The Kaplan-Meier nonparametric product limit method for censored data was used to estimate PFS.
Time Frame: Up to approximately 55 months
Population: All randomized participants analyzed in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chemoradiotherapy + Pembrolizumab | Chemoradiotherapy + Placebo for Pembrolizumab
Number analyzed (Participants) | 529 | 531
Months | 47.6 [47.6 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 47.5 [41.0 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Chemoradiotherapy + Pembrolizumab vs Chemoradiotherapy + Placebo for Pembrolizumab; Test type: Superiority; p = 0.0004, Log Rank — One sided p-value; Stratified by planned type of external beam radiation therapy (EBRT), stage at screening, and planned total radiotherapy dose; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.59 to 0.87] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate

2. Primary Outcome: Overall Survival (OS)
Description: OS is the time from randomization to death due to any cause. The Kaplan-Meier nonparametric product limit method for censored data was used to estimate OS.
Time Frame: Up to approximately 55 months
Population: All randomized participants analyzed in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chemoradiotherapy + Pembrolizumab | Chemoradiotherapy + Placebo for Pembrolizumab
Number analyzed (Participants) | 529 | 531
Months | NA [NA to NA] — NA = Median, upper and lower limits not reached at time of data cut-off due to insufficient number of participants with an event. | NA [NA to NA] — NA = Median, upper and lower limits not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Chemoradiotherapy + Pembrolizumab vs Chemoradiotherapy + Placebo for Pembrolizumab; Test type: Superiority; p = 0.0076, Log Rank — One sided p-value; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.57 to 0.94] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate

3. Secondary Outcome: PFS Per RECIST 1.1 as Assessed by Blinded Independent Central Review (BICR)
Description: PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. Unequivocal progression of non-target lesions is also considered PD. The Kaplan-Meier nonparametric product limit method for censored data was used to estimate PFS.
Time Frame: Up to approximately 55 months
Population: All randomized participants analyzed in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chemoradiotherapy + Pembrolizumab | Chemoradiotherapy + Placebo for Pembrolizumab
Number analyzed (Participants) | 529 | 531
Months | 48.9 [48.9 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [46.8 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Chemoradiotherapy + Pembrolizumab vs Chemoradiotherapy + Placebo for Pembrolizumab; Test type: Superiority; p = 0.0011, Log Rank — One-sided p-value; Stratified by planned type of EBRT, stage at screening, and planned total radiotherapy dose; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.58 to 0.89] — Based on Cox regression model with Efron's method of tie handling

4. Secondary Outcome: PFS Per RECIST 1.1 at Month 24 as Assessed by the Investigator
Description: PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, or by histopathologic confirmation of suspected disease progression, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. Unequivocal progression of non-target lesions is also considered PD. The percentage of participants with PFS as assessed by the investigator is presented.
Time Frame: 24 months
Population: All randomized participants analyzed in the treatment group to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Chemoradiotherapy + Pembrolizumab | Chemoradiotherapy + Placebo for Pembrolizumab
Number analyzed (Participants) | 529 | 531
Percentage of Participants | 70.6 [66.4 to 74.3] | 59.7 [55.3 to 63.8]
Statistical Analysis 1: Comparison: Chemoradiotherapy + Pembrolizumab vs Chemoradiotherapy + Placebo for Pembrolizumab; Test type: Other; Difference in Survival Rate = 10.9, 95% CI 2-sided [5.1 to 16.7] — Pembrolizumab minus Placebo

5. Secondary Outcome: PFS Per RECIST 1.1 at Month 24 as Assessed by BICR
Description: PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. Unequivocal progression of non-target lesions is also considered PD. The percentage of participants with PFS as assessed by BICR is presented.
Time Frame: 24 months
Population: All randomized participants analyzed in the treatment group to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Chemoradiotherapy + Pembrolizumab | Chemoradiotherapy + Placebo for Pembrolizumab
Number analyzed (Participants) | 529 | 531
Percentage of Participants | 76.0 [72.0 to 79.5] | 68.1 [63.8 to 72.0]
Statistical Analysis 1: Comparison: Chemoradiotherapy + Pembrolizumab vs Chemoradiotherapy + Placebo for Pembrolizumab; Test type: Other; Difference in Survival Rate = 7.9, 95% CI 2-sided [2.3 to 13.5] — Pembrolizumab minus Placebo

6. Secondary Outcome: Overall Survival (OS) at Month 36
Description: OS is the time from randomization to death due to any cause. The analysis was performed via Kaplan-Meier approach to estimate the OS rate at Month 36. The percentage of participants with OS at Month 36 is presented.
Time Frame: 36 months
Population: All randomized participants analyzed in the treatment group to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Chemoradiotherapy + Pembrolizumab | Chemoradiotherapy + Placebo for Pembrolizumab
Number analyzed (Participants) | 529 | 531
Percentage of Participants | 81.8 [78.1 to 84.9] | 74.4 [70.3 to 78.0]
Statistical Analysis 1: Comparison: Chemoradiotherapy + Pembrolizumab vs Chemoradiotherapy + Placebo for Pembrolizumab; Test type: Other; Difference in Survival Rate = 7.4, 95% CI 2-sided [2.3 to 12.5] — Pembrolizumab minus Placebo

7. Secondary Outcome: Complete Response (CR) Rate Per RECIST 1.1 at Week 12 as Assessed by the Investigator
Description: For participants who demonstrated a confirmed Complete Response (CR: Disappearance of all target and non-target lesions and also includes reduction of all nodal lesions to <10mm) per RECIST 1.1, CR rate is defined as the percentage of participants who experienced a CR. The percentage of participants with CR per RECIST 1.1 as assessed by the investigator at Week 12 is presented.
Time Frame: 12 weeks
Population: All randomized participants analyzed in the treatment group to which they were randomized. Participants with measurable disease at baseline. As the BICR and Investigator each measure and collect results differently, this can result in different numbers of participants with measurable disease at baseline, and hence different numbers analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Chemoradiotherapy + Pembrolizumab | Chemoradiotherapy + Placebo for Pembrolizumab
Number analyzed (Participants) | 521 | 522
Percentage of participants | 36.9 [32.7 to 41.2] | 33.5 [29.5 to 37.8]
Statistical Analysis 1: Comparison: Chemoradiotherapy + Pembrolizumab vs Chemoradiotherapy + Placebo for Pembrolizumab; Test type: Other; p = 0.1307, One-sided p-value for testing; Difference in Percentage = 3.3, 95% CI 2-sided [-2.5 to 9.1] — Pembrolizumab minus Placebo; Miettinen & Nurminen method stratified by planned type of EBRT, Stage at screening and planned total radiotherapy dose

8. Secondary Outcome: CR Rate Per RECIST 1.1 at Week 12 as Assessed by BICR
Description: For participants who demonstrated a confirmed CR: Disappearance of all target and non-target lesions and also includes reduction of all nodal lesions to <10mm) per RECIST 1.1, CR rate is defined as the percentage of participants who experienced a CR. The percentage of participants with CR per RECIST 1.1 as assessed by BICR at Week 12 is presented.
Time Frame: 12 weeks
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Chemoradiotherapy + Pembrolizumab | Chemoradiotherapy + Placebo for Pembrolizumab
Number analyzed (Participants) | 527 | 531
Percentage of participants | 42.9 [38.6 to 47.2] | 42.2 [37.9 to 46.9]
Statistical Analysis 1: Comparison: Chemoradiotherapy + Pembrolizumab vs Chemoradiotherapy + Placebo for Pembrolizumab; Test type: Other; p = 0.4082, One-sided p-value for testing; Difference in Percentage = 0.7, 95% CI 2-sided [-5.2 to 6.7] — Pembrolizumab minus Placebo; Miettinen & Nurminen method stratified by planned type of EBRT, Stage at screening and planned total radiotherapy dose

9. Secondary Outcome: Objective Response Rate (ORR) Per RECIST 1.1 as Assessed by the Investigator
Description: ORR is defined as the percentage of participants who have a Complete Response (CR: Disappearance of all target and non-target lesions and also includes reduction of all nodal lesions to <10mm) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions and includes no unequivocal progression in non-target lesions) per RECIST 1.1.
Time Frame: Up to approximately 55 months
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Chemoradiotherapy + Pembrolizumab | Chemoradiotherapy + Placebo for Pembrolizumab
Number analyzed (Participants) | 521 | 522
Percentage of participants | 87.3 [84.2 to 90.1] | 83.7 [80.3 to 86.8]
Statistical Analysis 1: Comparison: Chemoradiotherapy + Pembrolizumab vs Chemoradiotherapy + Placebo for Pembrolizumab; Test type: Other; p = 0.0496, One-sided p-value for testing; Difference in Percentage = 3.6, 95% CI 2-sided [-0.7 to 7.9] — Pembrolizumab minus Placebo; Miettinen & Nurminen method stratified by planned type of EBRT, Stage at screening and planned total radiotherapy dose

10. Secondary Outcome: ORR Per RECIST 1.1 as Assessed by BICR
Description: as for outcome 9
Time Frame: Up to approximately 55 months
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Chemoradiotherapy + Pembrolizumab | Chemoradiotherapy + Placebo for Pembrolizumab
Number analyzed (Participants) | 527 | 531
Percentage of participants | 90.5 [87.7 to 92.9] | 88.3 [85.3 to 90.9]
Statistical Analysis 1: Comparison: Chemoradiotherapy + Pembrolizumab vs Chemoradiotherapy + Placebo for Pembrolizumab; Test type: Other; p = 0.1244, One-sided p-value for testing; Difference in Percentage = 2.2, 95% CI 2-sided [-1.5 to 5.9] — Pembrolizumab minus Placebo; Miettinen & Nurminen method stratified by planned type of EBRT, Stage at screening and planned total radiotherapy dose

11. Secondary Outcome: PFS Per RECIST 1.1 in Programmed Cell Death 1 Ligand 1 (PD-L1) Positive Participants as Assessed by the Investigator
Description: PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, or by histopathologic confirmation of suspected disease progression, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. Unequivocal progression of non-target lesions is also considered PD. PD-L1 positive participants have a combined positivity score (CPS) equal or greater than 1. The Kaplan-Meier nonparametric product limit method for censored data was used to estimate PFS.
Time Frame: Up to approximately 55 months
Population: All randomized participants analyzed in the treatment group to which they were randomized. PD-L1 positive participants were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chemoradiotherapy + Pembrolizumab | Chemoradiotherapy + Placebo for Pembrolizumab
Number analyzed (Participants) | 502 | 498
Months | 47.6 [47.6 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 47.5 [41.0 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Chemoradiotherapy + Pembrolizumab vs Chemoradiotherapy + Placebo for Pembrolizumab; Test type: Other; p = 0.0010, Log Rank — One-sided p-value; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.59 to 0.89] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate

12. Secondary Outcome: PFS Per RECIST 1.1 in PD-L1 Positive Participants as Assessed by BICR
Description: PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. Unequivocal progression of non-target lesions is also considered PD. PD-L1 positive participants have a CPS equal or greater than 1. The Kaplan-Meier nonparametric product limit method for censored data was used to estimate PFS.
Time Frame: Up to approximately 55 months
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chemoradiotherapy + Pembrolizumab | Chemoradiotherapy + Placebo for Pembrolizumab
Number analyzed (Participants) | 502 | 498
Months | 48.9 [48.9 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [46.8 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Chemoradiotherapy + Pembrolizumab vs Chemoradiotherapy + Placebo for Pembrolizumab; Test type: Other; p = 0.0016, Log Rank — One-sided p-value; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.58 to 0.90] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate

13. Secondary Outcome: OS in PD-L1 Positive Participants
Description: OS is the time from randomization to death due to any cause. PD-L1 positive participants have a CPS equal or greater than 1. The Kaplan-Meier nonparametric product limit method for censored data was used to estimate OS.
Time Frame: Up to approximately 55 months
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chemoradiotherapy + Pembrolizumab | Chemoradiotherapy + Placebo for Pembrolizumab
Number analyzed (Participants) | 502 | 498
Months | NA [NA to NA] — NA = Median, upper and lower limits not reached at time of data cut-off due to insufficient number of participants with an event. | NA [NA to NA] — NA = Median, upper and lower limits not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Chemoradiotherapy + Pembrolizumab vs Chemoradiotherapy + Placebo for Pembrolizumab; Test type: Other; p = 0.0083, Log Rank — One-sided p-value; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.56 to 0.95] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate

14. Secondary Outcome: PFS After Next-Line Treatment (PFS 2) Following Discontinuation of Study Treatment
Description: PFS is defined as the time from randomization to the first documented progressive disease (PD) on next-line treatment or death due to any cause, whichever occurs first, as assessed by the investigator. PFS 2 is measured after next-line treatment following discontinuation of study treatment administration.
Time Frame: Up to approximately 55 months
Population: All randomized participants analyzed in the treatment group to which they were randomized
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chemoradiotherapy + Pembrolizumab | Chemoradiotherapy + Placebo for Pembrolizumab
Number analyzed (Participants) | 529 | 531
Months | NA [NA to NA] — NA = Median, upper and lower limits not reached at time of data cut-off due to insufficient number of participants with an event. | NA [NA to NA] — NA = Median, upper and lower limits not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Chemoradiotherapy + Pembrolizumab vs Chemoradiotherapy + Placebo for Pembrolizumab; Test type: Other; p = 0.0015, Log Rank — One-sided p-value; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.54 to 0.88] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate

15. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Global Health Status Score
Description: The EORTC QLQ-C30 is a questionnaire that rates the overall quality of life in cancer participants. The first 28 questions use a 4-point scale (1=not at all to 4=very much) for evaluating function (physical, role, social, cognitive, emotional), symptoms (diarrhea, fatigue, dyspnea, appetite loss, insomnia, nausea/vomiting, constipation, and pain) and financial difficulties. The last 2 questions use a 7-point scale (1=very poor to 7=excellent) to evaluate overall health and quality of life. Global scores are converted to a score of 0 to 100, with a higher score indicating improved health status. The change from baseline in EORTC QLQ-C30 score will be presented.
Time Frame: Baseline and week 36
Population: Randomized participants who have at least 1 patient reported outcome (PRO) assessment for QLQ-C30 available and have received at least 1 dose of study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Chemoradiotherapy + Pembrolizumab | Chemoradiotherapy + Placebo for Pembrolizumab
Number analyzed (Participants) | 503 | 506
Score on a scale | 7.51 [5.30 to 9.73] | 7.44 [5.23 to 9.66]
Statistical Analysis 1: Comparison: Chemoradiotherapy + Pembrolizumab vs Chemoradiotherapy + Placebo for Pembrolizumab; Test type: Other; p = 0.9593, cLDA model; Difference LS Means = 0.07, 95% CI 2-sided [-2.66 to 2.80] — Pembrolizumab minus placebo; Based on a cLDA model with the patient-reported outcome (PRO) scores as the response variable with covariates for treatment by study visit interaction, and stratified by planned type of EBRT

16. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Physical Function Score
Description: The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=not at all to 4=very much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better quality of life. The change from baseline in physical function (EORTC QLQ-C30 Items 1-5) score will be presented.
Time Frame: Baseline and week 36
Population: Randomized participants who have at least 1 PRO assessment for QLQ-C30 available and have received at least 1 dose of study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Chemoradiotherapy + Pembrolizumab | Chemoradiotherapy + Placebo for Pembrolizumab
Number analyzed (Participants) | 503 | 506
Score on a scale | 2.74 [1.16 to 4.33] | 2.07 [0.48 to 3.65]
Statistical Analysis 1: Comparison: Chemoradiotherapy + Pembrolizumab vs Chemoradiotherapy + Placebo for Pembrolizumab; Test type: Other; p = 0.5145, cLDA model; Difference LS Means = 0.68, 95% CI 2-sided [-1.36 to 2.71] — Pembrolizumab minus placebo; Based on a cLDA model with the PRO scores as the response variable with covariates for treatment by study visit interaction, and stratified by planned type of EBRT

17. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Symptom Specific Scale for Cervical Cancer (EORTC QLQ-CX24) Score
Description: The EORTC QLQ-CX24 is a questionnaire that rates the symptoms common to women with cervical cancer and evaluates the impact of disease and/or treatments. The 24 items use a 4-point scale (1=not at all to 4=very much) and are classified into 3 multi-item scales, 11 items with symptom experience, 3 items with body image, and 4 items with sexual/ vaginal functioning. The other items of the questionnaire are lymphedema, peripheral neuropathy, menopausal symptom, sexual worry, sexual activity, and sexual enjoyment. Total scores are linearly transformed and range from 0 (no symptoms) to 100 (most severe symptoms). The change from baseline in EORTC QLQ-CX24 score is presented, with negative scores representing an improvement from baseline and vice versa.
Time Frame: Baseline and Week 36
Population: Randomized participants who have at least 1 PRO assessment for QLQ-CX24 available and have received at least 1 dose of study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Chemoradiotherapy + Pembrolizumab | Chemoradiotherapy + Placebo for Pembrolizumab
Number analyzed (Participants) | 503 | 504
Score on a scale | -8.86 [-10.03 to -7.69] | -9.60 [-10.78 to -8.43]
Statistical Analysis 1: Comparison: Chemoradiotherapy + Pembrolizumab vs Chemoradiotherapy + Placebo for Pembrolizumab; Test type: Other; p = 0.2953, cLDA model; Difference LS Means = 0.75, 95% CI 2-sided [-0.65 to 2.15] — Pembrolizumab minus placebo; [other analysis details as in outcome 16, analysis 1]

18. Secondary Outcome: Number of Participants Who Experience One or More Adverse Events (AEs)
Description: An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.
Time Frame: Up to 55 months
Population: All randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemoradiotherapy + Pembrolizumab | Chemoradiotherapy + Placebo for Pembrolizumab
Number analyzed (Participants) | 528 | 530
Participants | 528 | 526

19. Secondary Outcome: Number of Participants Who Discontinue Study Treatment Due to an AE
Description: as for outcome 18
Time Frame: Up to 32 months
Population: All randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemoradiotherapy + Pembrolizumab | Chemoradiotherapy + Placebo for Pembrolizumab
Number analyzed (Participants) | 528 | 530
Participants | 112 | 79

ADVERSE EVENTS:
Time Frame: All-cause mortality (ACM): from allocation up to a maximum of 55 months. Adverse events (AEs): from start of treatment up to a maximum of 55 months.
Description: The ACM population were allocated participants; the AE population were treated participants. As it was pre-specified that disease progression of cancer was not considered an AE unless related to study drug, the following AE preferred terms not related to the drug were excluded: Neoplasm progression, Malignant neoplasm progression and Disease progression.
Groups:
- Pembrolizumab + CCRT: Participants received pembrolizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle (Q3W) for 5 cycles followed by pembrolizumab 400 mg IV on Day 1 of each 6-week cycle (Q6W) for an additional 15 cycles. During the Q3W dosing period of pembrolizumab, participants received concurrent chemoradiotherapy. The standard of care chemoradiotherapy regimen includes cisplatin 40 mg/m^2 IV once per week (QW) for 5 or 6 weeks plus external beam radiotherapy (EBRT) followed by brachytherapy with minimum total radiotherapy dose of 80 Gray Units (Gy) for volume-directed and 75 Gy for point-directed given with the total duration of radiation treatment not to exceed 50 days (with an extension to a maximum of 56 days for unforeseen delays).
- Placebo + CCRT: Participants received placebo for pembrolizumab IV on Day 1 of each 3-week cycle (Q3W) for 5 cycles followed by placebo IV on Day 1 of each 6-week cycle (Q6W) for an additional 15 cycles. During the Q3W dosing period of placebo, participants received concurrent chemoradiotherapy. The standard of care chemoradiotherapy regimen includes cisplatin 40 mg/m^2 IV once per week (QW) for 5 or 6 weeks plus external beam radiotherapy (EBRT) followed by brachytherapy with minimum total radiotherapy dose of 80 Gray Units (Gy) for volume-directed and 75 Gy for point-directed given with the total duration of radiation treatment not to exceed 50 days (with an extension to a maximum of 56 days for unforeseen delays).
Arm/Group | Pembrolizumab + CCRT | Placebo + CCRT
All-Cause Mortality (participants affected / at risk) | 107/529 | 140/531
Serious Adverse Events (participants affected / at risk) | 175/528 | 153/530
Other Adverse Events (participants affected / at risk) | 528/528 | 525/530
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + CCRT (N=528) | Placebo + CCRT (N=530)
Anaemia (Blood and lymphatic system disorders) | 16 (20) | 13 (13)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 4 (4)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 0 (0)
Glucocorticoid deficiency (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Secondary adrenocortical insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (5)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Autoimmune colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 3 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 10 (11) | 6 (7)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Haemoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Immune-mediated gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2)
Intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 5 (5)
Neutropenic colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (5)
Death (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 2 (2)
Hyperpyrexia (General disorders) | 1 (1) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 14 (16) | 10 (12)
Ulcer (General disorders) | 1 (1) | 0 (0)
Acute cholecystitis necrotic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Appendiceal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 4 (5)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 2 (2)
Infection (Infections and infestations) | 2 (2) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Intrauterine infection (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 2 (2) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lymphangitis (Infections and infestations) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pelvic abscess (Infections and infestations) | 1 (1) | 0 (0)
Pelvic infection (Infections and infestations) | 2 (2) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Psoas abscess (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 6 (7) | 6 (6)
Pyelonephritis acute (Infections and infestations) | 2 (2) | 0 (0)
Pyometra (Infections and infestations) | 3 (3) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 6 (6) | 5 (6)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Toxic shock syndrome streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 18 (24) | 13 (16)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 4 (4) | 1 (1)
Uterine infection (Infections and infestations) | 2 (3) | 0 (0)
Vaginal infection (Infections and infestations) | 2 (2) | 1 (1)
Vulvitis (Infections and infestations) | 2 (2) | 0 (0)
Vulvovaginitis (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Cystitis radiation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 5 (6) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural headache (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation proctitis (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (3)
Urostomy complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Uterine perforation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 0 (0)
Blood corticotrophin decreased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1)
Blood magnesium decreased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 2 (2)
Platelet count decreased (Investigations) | 4 (4) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Appendix cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Intracranial mass (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 3 (3) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 1 (2)
Device occlusion (Product Issues) | 1 (1) | 2 (2)
Stent malfunction (Product Issues) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 6 (9)
Autoimmune nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 6 (6) | 3 (3)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteral cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric dilatation (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary tract disorder (Renal and urinary disorders) | 1 (2) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2) | 1 (1)
Urogenital fistula (Renal and urinary disorders) | 1 (1) | 1 (1)
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Uterine fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 6 (7) | 5 (6)
Vaginal perforation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulval disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 4 (4)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + CCRT (N=528) | Placebo + CCRT (N=530)
Anaemia (Blood and lymphatic system disorders) | 356 (549) | 342 (489)
Leukopenia (Blood and lymphatic system disorders) | 129 (216) | 97 (160)
Lymphopenia (Blood and lymphatic system disorders) | 52 (77) | 56 (80)
Neutropenia (Blood and lymphatic system disorders) | 124 (200) | 107 (161)
Thrombocytopenia (Blood and lymphatic system disorders) | 80 (89) | 69 (86)
Tinnitus (Ear and labyrinth disorders) | 31 (32) | 35 (39)
Hyperthyroidism (Endocrine disorders) | 62 (70) | 15 (15)
Hypothyroidism (Endocrine disorders) | 119 (146) | 39 (48)
Abdominal pain (Gastrointestinal disorders) | 78 (94) | 78 (102)
Abdominal pain upper (Gastrointestinal disorders) | 35 (39) | 35 (39)
Constipation (Gastrointestinal disorders) | 118 (139) | 122 (151)
Diarrhoea (Gastrointestinal disorders) | 297 (479) | 296 (421)
Dyspepsia (Gastrointestinal disorders) | 21 (21) | 30 (33)
Nausea (Gastrointestinal disorders) | 318 (442) | 337 (460)
Vomiting (Gastrointestinal disorders) | 158 (237) | 177 (267)
Asthenia (General disorders) | 92 (119) | 75 (98)
Fatigue (General disorders) | 103 (124) | 114 (128)
Malaise (General disorders) | 22 (24) | 29 (34)
Pyrexia (General disorders) | 78 (112) | 76 (100)
COVID-19 (Infections and infestations) | 59 (62) | 52 (57)
Cystitis (Infections and infestations) | 38 (41) | 26 (29)
Urinary tract infection (Infections and infestations) | 113 (182) | 145 (224)
Radiation skin injury (Injury, poisoning and procedural complications) | 34 (34) | 32 (34)
Alanine aminotransferase increased (Investigations) | 116 (170) | 87 (116)
Aspartate aminotransferase increased (Investigations) | 111 (148) | 72 (99)
Blood alkaline phosphatase increased (Investigations) | 44 (57) | 38 (50)
Blood creatinine increased (Investigations) | 60 (100) | 64 (103)
Blood lactate dehydrogenase increased (Investigations) | 27 (31) | 15 (20)
Lymphocyte count decreased (Investigations) | 80 (120) | 94 (147)
Neutrophil count decreased (Investigations) | 164 (380) | 151 (355)
Platelet count decreased (Investigations) | 117 (164) | 112 (154)
SARS-CoV-2 test positive (Investigations) | 34 (34) | 31 (32)
Weight decreased (Investigations) | 82 (91) | 81 (88)
White blood cell count decreased (Investigations) | 175 (518) | 187 (554)
Decreased appetite (Metabolism and nutrition disorders) | 95 (106) | 106 (115)
Hyperglycaemia (Metabolism and nutrition disorders) | 45 (68) | 44 (58)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 40 (49) | 38 (48)
Hypocalcaemia (Metabolism and nutrition disorders) | 35 (46) | 36 (44)
Hypokalaemia (Metabolism and nutrition disorders) | 114 (176) | 92 (133)
Hypomagnesaemia (Metabolism and nutrition disorders) | 129 (170) | 124 (161)
Hyponatraemia (Metabolism and nutrition disorders) | 59 (74) | 57 (68)
Arthralgia (Musculoskeletal and connective tissue disorders) | 62 (75) | 67 (90)
Back pain (Musculoskeletal and connective tissue disorders) | 46 (51) | 60 (73)
Myalgia (Musculoskeletal and connective tissue disorders) | 31 (36) | 38 (41)
Dizziness (Nervous system disorders) | 30 (30) | 46 (55)
Dysgeusia (Nervous system disorders) | 25 (26) | 28 (30)
Headache (Nervous system disorders) | 67 (84) | 72 (101)
Insomnia (Psychiatric disorders) | 50 (58) | 49 (57)
Dysuria (Renal and urinary disorders) | 78 (92) | 73 (86)
Haematuria (Renal and urinary disorders) | 29 (34) | 26 (35)
Proteinuria (Renal and urinary disorders) | 27 (31) | 18 (21)
Pelvic pain (Reproductive system and breast disorders) | 52 (58) | 65 (77)
Vaginal discharge (Reproductive system and breast disorders) | 30 (34) | 36 (42)
Vaginal haemorrhage (Reproductive system and breast disorders) | 36 (41) | 44 (53)
Cough (Respiratory, thoracic and mediastinal disorders) | 31 (34) | 29 (32)
Pruritus (Skin and subcutaneous tissue disorders) | 36 (43) | 31 (31)
Rash (Skin and subcutaneous tissue disorders) | 47 (54) | 25 (39)
Hot flush (Vascular disorders) | 26 (27) | 49 (51)
Hypertension (Vascular disorders) | 31 (37) | 16 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/45/NCT04221945/Prot_SAP_000.pdf